CLINICAL TRIAL: NCT02967523
Title: Surefire Precision Infusion System Registry
Status: Terminated | Type: Observational
Sponsor: Surefire Medical, Inc. (Industry)
Responsible Party: Sponsor
Organization: SurefireMedical (Unknown)
Other Study IDs: 26 October 2016
Record Dates: First submitted 2016-11-16; First posted 2016-11-18 (Estimated); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma; DEB-TACE
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: DEB-TACE with Surefire Precision Infusion System — Subjects have undergone/will undergo DEB-TACE using the Surefire Precision Infusion System.

SUMMARY:
This project involves the collection and analysis of retrospective and prospective data on patients diagnosed with hepatocellular carcinoma (HCC) in which the Surefire Precision Infusion System was used/will used be to deliver transarterial chemoembolization with doxorubicin-eluting beads (DEB-TACE). The purpose is to compare tumor and medical response in a real-world setting as well as identify potential areas for future clinical research.

DETAILED DESCRIPTION:
Conventional transarterial chemoembolization with lipiodol/doxorubicin (cTACE) is known to prolong survival compared to supportive therapy in certain patients with unresectable HCC, including patients with unilateral portal vein invasion (PVI). The best results for cTACE occur when the dose is delivered in a highly targeted manner into the tumor. Dense accumulation of embolic spheres or lipiodol into the tumor as documented by computed tomography (CT) has been shown to have improved outcomes. However, with standard endhole catheters, achieving maximum delivery of embolic agents is significantly limited by the development of stasis, non-target delivery and subsequent non-target injury. Thus, when this procedure is performed with endhole catheters, there is significant variability in the delivery of the agent that is entirely dependent on the flow pattern of the target tumor. Therefore, current techniques result in various degrees of embolization with variability in dosages and angiographic endpoints.

DEB-TACE is a relatively new modality associated with favorable systemic doxorubicin exposure/toxicity and liver-specific toxicity compared to cTACE. It is currently utilized for: (1) patients who have unresectable HCC; (2) patients who meet the Milan Criteria and are currently on liver transplantation lists; and (3) downstaging patients into Milan Criteria for possible liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone or will undergo DEB-TACE for HCC delivered by the Surefire® Precision Infusion System
* Patients aged 18 years or older
* Diagnosis of HCC
* Has a discrete hepatic artery(s) feeding the vessel with diameter(s) of the vessels ≥ 1.5 mm

Exclusion Criteria:

* Contraindications for doxorubicin administration
* Vessels providing flow to the tumor that are < 1.5 mm in diameter(s)
* Patients who are unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have been diagnosed with HCC in which the Surefire Precision Infusion System was used/will be used to deliver DEB-TACE.
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2016-05; Primary Completion 2018-06-18 (Actual); Study Completion 2018-06-18 (Actual)

PRIMARY OUTCOMES:
Objective tumor response | 6 months following initial DEB-TACE procedure.

SECONDARY OUTCOMES:
Objective tumor response | 1 and 3 months following initial DEB-TACE procedure
Dose of doxorubicin-eluting beads used during DEB-TACE procedure(s) | 6 months following initial DEB-TACE procedure
Tumor characteristics | DEB-TACE procedure(s)
  Number of lesions, location of lesions (uni-lobar versus bi-lobar), and distribution (unifocal, multi-focal, diffuse)
Size of doxorubicin-eluting beads used during DEB-TACE procedure(s) | DEB-TACE procedure(s)
Changes in alpha-fetoprotein (AFP) blood levels | 1, 3 and 6 months following initial DEB-TACE procedure

CONTACTS AND LOCATIONS:
Overall Officials: Baljendra Kapoor, MD, Principal Investigator — The Cleveland Clinic
Locations (10):
- United States (10):
  - UCLA, Los Angeles, California
  - USC, Los Angeles, California
  - UCSD, San Diego, California
  - Medstar Georgetown University Hospital, Washington D.C., District of Columbia
  - Florida Hospital, Orlando, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - University of Maryland Medical Center, Baltimore, Maryland
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No